CLINICAL TRIAL: NCT04608344
Title: A Phase 1 Study to Evaluate OATP Transporter-Mediated Drug-Drug Interactions Between Filgotinib and Statins as Probe Drugs in Healthy Participants
Brief Title: Study to Evaluate Organic Anion Transporting Polypeptide (OATP) Transporter-Mediated Drug-Drug Interactions Between Filgotinib and Statins as Probe Drugs in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Collaborators: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: GS-US-417-5937
Record Dates: First submitted 2020-10-23; First posted 2020-10-29 (Actual); Results first posted 2022-01-19 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-05

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Atorvastatin; Pravastatin; Rosuvastatin Calcium; GLPG0634

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sequence AB (Experimental): Participants will receive atorvastatin (ATV) 40 mg tablet on Day 1, followed by a washout period of 1 day, and then pravastatin (PRA) 40 mg + rosuvastatin (ROS) 10 mg tablets on Day 3 in Treatment A, Period 1. In Treatment B, Period 2 participants will receive filgotinib 200 mg tablet once daily for 11 days, with ATV 40 mg on Day 12 and PRA 40 mg + ROS 10 mg tablets on Day 14. Period 1 and Period 2 will be separated by a washout period of 3 days.
  Interventions: Drug: Atorvastatin; Drug: Pravastatin; Drug: Rosuvastatin; Drug: Filgotinib
- Sequence BA (Experimental): Participants will receive filgotinib 200 mg tablet once daily for 11 days, with ATV 40 mg on Day 6 and PRA 40 mg + ROS 10 mg tablets on Day 8 in Treatment B, Period 1. In Treatment A, Period 2 participants will receive ATV 40 mg tablet on Day 18, followed by a washout period of 1 day and PRA 40 mg + ROS 10 mg tablets on Day 20. Period 1 and Period 2 will be separated by a washout period of 6 days.
  Interventions: Drug: Atorvastatin; Drug: Pravastatin; Drug: Rosuvastatin; Drug: Filgotinib

INTERVENTIONS:
Drug: Atorvastatin — Administered as single dose tablet orally.
Drug: Pravastatin — Administered as single dose tablet orally.
Drug: Rosuvastatin — Administered as single dose tablet orally.
Drug: Filgotinib — Administered as tablet orally once daily for 11 days.
  Other Names: GS-6034; GLPG0634; Jyseleca

SUMMARY:
The primary objective of this study is to evaluate the effect of filgotinib on a mixed organic anion transporting polypeptide/cytochrome P450 3A (OATP/CYP3A), OATP/ breast cancer resistance protein (BCRP), and OATP substrates using phenotypic probes.

ELIGIBILITY:
Key Inclusion Criteria:

* Be a nonsmoker. The use of nicotine or nicotine-containing products must be discontinued 90 days prior to the first dose of study drug.
* Have a calculated body mass index (BMI) of greater than or equal to (≥) 19.0 and less than or equal to (≤) 30.0 kilogram per meter square (kg/m^2) at screening.
* Have a creatinine clearance (CLcr) ≥ 90 milliliters per minute (mL/min) (using the Cockcroft-Gault method) based on serum creatinine and actual body weight as measured at screening and upon admission.
* Female participants of childbearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test at clinic admission.
* Male participants must be surgically sterile.
* Male participants and female participants of childbearing potential who engage in heterosexual intercourse must agree to use protocol-specified method(s) of contraception.
* Screening laboratory evaluations and 12-lead electrocardiogram (ECG) evaluations must be without clinically significant abnormalities as assessed by the investigator.
* Have liver biometric tests such as alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase, and total bilirubin below the upper limit of normal at screening.
* Must be willing and able to comply with all study requirements.
* Must, in the opinion of the investigator, be in good health based upon medical history and physical examination, including vital signs.
* Participants must not have donated blood within 56 days of study entry or plasma within 7 days of study entry and must refrain from blood donation from clinic admission, throughout the study period, and continuing for at least 30 days following the last dose of study drug.

Key Exclusion Criteria:

* Positive serum pregnancy test (Female participants).
* Lactating female.
* Have received any investigational drug/device within 30 days prior to study dosing (or within 5 half-lives of the drug, whichever is longer).
* Have current alcohol or substance abuse judged by the investigator to potentially interfere with participant compliance or participant safety, or a positive drug or alcohol test at screening or admission.
* Have a positive test result for human immunodeficiency virus type 1 (HIV-1) antibody, hepatitis B virus (HBV) surface antigen (HBsAg), or hepatitis C virus (HCV) antibody at screening.
* Have positive Coronavirus Disease 2019 (COVID-19) Real-Time Reverse.
* Transcriptase-Polymerase Chain Reaction (RT-PCR) testing on screening and admission.
* Have poor venous access that limits phlebotomy.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2021-01-13 (Actual); Study Completion 2021-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (1):
- Prism Research, LLC, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gileadclinicaltrials.com/transparency-policy/
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gileadclinicaltrials.com/transparency-policy/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at a study site in the United States. The first participant was screened on 04 November 2020. The last study visit occurred on 13 January 2021.
Pre-assignment Details: 55 participants were screened.
Groups:
- Sequence AB: Participants received a single oral dose of atorvastatin (ATV) 40 mg tablet on Day 1, followed by a washout period of 1 day, and then a single oral dose of pravastatin (PRA) 40 mg + rosuvastatin (ROS) 10 mg tablets on Day 3 in Treatment A, Period 1. In Treatment B, Period 2 participants received an oral dose of filgotinib 200 mg tablet once daily for 11 days, with a single oral dose of ATV 40 mg on Day 12 and a single oral dose of PRA 40 mg + ROS 10 mg tablets on Day 14. Period 1 and Period 2 were separated by a washout period of 3 days.
- Sequence BA: Participants received an oral dose of filgotinib 200 mg tablet once daily for 11 days, with a single oral dose of ATV 40 mg on Day 6 and a single oral dose of PRA 40 mg + ROS 10 mg tablets on Day 8 in Treatment B, Period 1. In Treatment A, Period 2 participants received single oral dose of ATV 40 mg tablet on Day 18, followed by a washout period of 1 day and a single oral dose of PRA 40 mg + ROS 10 mg tablets on Day 20. Period 1 and Period 2 were separated by a washout period of 6 days.
Period: Period 1 (AB: 3 Days, BA: 11 Days)
Arm/Group | Sequence AB | Sequence BA
Started | 14 | 13
Completed | 13 | 12
Not Completed | 1 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Investigator's Discretion | 1 | 0
Period: Period 2 (AB: 11 Days, BA: 3 Days)
Arm/Group | Sequence AB | Sequence BA
Started | 13 | 12
Completed | 13 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all randomized participants who received at least 1 dose of any study drug.
Groups:
- Sequence AB: Participants received a single oral dose of ATV 40 mg tablet on Day 1, followed by a washout period of 1 day, and then a single oral dose of PRA 40 mg + ROS 10 mg tablets on Day 3 in Treatment A, Period 1. In Treatment B, Period 2 participants received an oral dose of filgotinib 200 mg tablet once daily for 11 days, with a single oral dose of ATV 40 mg on Day 12 and a single oral dose of PRA 40 mg + ROS 10 mg tablets on Day 14. Period 1 and Period 2 were separated by a washout period of 3 days.
- Total: Total of all reporting groups
Arm/Group | Sequence AB | Sequence BA | Total
Number analyzed (Participants) | 14 | 13 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (7.2) | 29 (7.6) | 30 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 12 | 26
  Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 14 | 12 | 26
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 10 | 9 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic (PK) Parameter: AUClast of ATV, PRA, and ROS
Description: AUClast is defined as the concentration of drug from time zero to the last observable concentration.
Time Frame: AB (Days 1,3,12,14) and BA (Days 6,8,18,20): Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48 postdose; AB (Days 1,12) and BA (Days 6,18): 5,10,36 hours post dose; AB (Days 3,14) and BA (Days 8,20): 72 hours postdose
Population: Participants in the PK Analysis Set (all randomized participants who received at least 1 dose of study drug and had at least 1 non-missing PK concentration datum reported by PK laboratory for each respective analyte) with available data were analyzed.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Groups:
- Atorvastatin: Participants either received a single oral dose of ATV 40 mg tablet on Day 1 in Treatment A, Period 1 or a single oral dose of ATV 40 mg on Day 12 in Treatment B, Period 2 or a single oral dose of ATV 40 mg on Day 6 in Treatment B, Period 1 or a single oral dose of ATV 40 mg tablet on Day 18 in Treatment A, Period 2.
- Pravastatin + Rosuvastatin: Participants either received a single oral dose of PRA 40 mg + ROS 10 mg tablets on Day 3 in Treatment A, Period 1 or a single oral dose of PRA 40 mg + ROS 10 mg tablets on Day 14 in Treatment B, Period 2 or a single oral dose of PRA 40 mg + ROS 10 mg tablets on Day 8 in Treatment B, Period 1 or a single oral dose of PRA 40 mg + ROS 10 mg tablets on Day 20 in Treatment A, Period 2.
- Filgotinib + Atorvastatin: Participants either received an oral dose of filgotinib 200 mg tablet once daily for 11 days, with a single oral dose of ATV 40 mg on Day 12 in Treatment B, Period 2 or an oral dose of filgotinib 200 mg tablet once daily for 11 days, with a single oral dose of ATV 40 mg on Day 6 in Treatment B, Period 1.
- Filgotinib + Pravastatin + Rosuvastatin: Participants either received an oral dose of filgotinib 200 mg tablet once daily for 11 days with a single oral dose of PRA 40 mg + ROS 10 mg tablets on Day 14 in Treatment B, Period 2 or an oral dose of filgotinib 200 mg tablet once daily for 11 days with a single oral dose of PRA 40 mg + ROS 10 mg tablets on Day 8 in Treatment B, Period 1.
Arm/Group | Atorvastatin | Pravastatin + Rosuvastatin | Filgotinib + Atorvastatin | Filgotinib + Pravastatin + Rosuvastatin
Number analyzed (Participants) | 25 | 25 | 26 | 26
h*ng/mL
  ATV: number analyzed (Participants) | 25 | 0 | 26 | 0
  ATV | 78.8 (39.10) |  | 70.2 (27.08) |
  PRA: number analyzed (Participants) | 0 | 25 | 0 | 26
  PRA |  | 199.5 (115.64) |  | 232.5 (137.76)
  ROS: number analyzed (Participants) | 0 | 25 | 0 | 26
  ROS |  | 62.6 (29.03) |  | 89.3 (34.63)

2. Primary Outcome: PK Parameter: AUCinf of ATV, PRA, and ROS
Description: AUCinf is defined as the concentration of drug extrapolated to infinite time.
Time Frame: as for outcome 1
Population: Participants in the PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Atorvastatin | Pravastatin + Rosuvastatin | Filgotinib + Atorvastatin | Filgotinib + Pravastatin + Rosuvastatin
Number analyzed (Participants) | 25 | 25 | 26 | 26
h*ng/mL
  ATV: number analyzed (Participants) | 25 | 0 | 26 | 0
  ATV | 80.8 (39.76) |  | 71.8 (27.30) |
  PRA: number analyzed (Participants) | 0 | 25 | 0 | 26
  PRA |  | 201.3 (116.38) |  | 234.8 (137.43)
  ROS: number analyzed (Participants) | 0 | 25 | 0 | 26
  ROS |  | 66.0 (29.53) |  | 92.3 (34.94)

3. Primary Outcome: PK Parameter: Cmax of ATV, PRA, and ROS
Description: Cmax is defined as the maximum observed concentration of drug.
Time Frame: as for outcome 1
Population: Participants in the PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Atorvastatin | Pravastatin + Rosuvastatin | Filgotinib + Atorvastatin | Filgotinib + Pravastatin + Rosuvastatin
Number analyzed (Participants) | 25 | 25 | 26 | 26
ng/mL
  ATV: number analyzed (Participants) | 25 | 0 | 26 | 0
  ATV | 19.7 (13.50) |  | 15.0 (7.81) |
  PRA: number analyzed (Participants) | 0 | 25 | 0 | 26
  PRA |  | 84.2 (56.60) |  | 99.2 (65.68)
  ROS: number analyzed (Participants) | 0 | 25 | 0 | 26
  ROS |  | 7.5 (4.17) |  | 12.3 (6.00)

4. Secondary Outcome: Percentage of Participants Experiencing Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant administered a study drug, which did not necessarily have a causal relationship with the treatment. AE was therefore any unfavorable and/or unintended sign, symptom, or disease temporally associated with the use of the study drug, whether or not considered related to the study drug. TEAEs: AE with an onset date on or after the study drug start date and no later than 30 days after study drug stop date; or any AE leading to study drug discontinuation.
Time Frame: Sequence AB: First dose up to 47 days, Sequence BA: First dose up to 50 days
Population: All randomized participants who received at least 1 dose of that particular study drug.
Measure: Number; unit: percentage of participants
Groups:
- Filgotinib: Participants either received an oral dose of filgotinib 200 mg tablet once daily for 11 days in Treatment B, Period 2 or an oral dose of filgotinib 200 mg tablet once daily for 11 days in Treatment B, Period 1.
Arm/Group | Atorvastatin | Pravastatin + Rosuvastatin | Filgotinib | Filgotinib + Atorvastatin | Filgotinib + Pravastatin + Rosuvastatin
Number analyzed (Participants) | 26 | 25 | 26 | 26 | 26
percentage of participants | 19.2 | 24.0 | 65.4 | 7.7 | 11.5

5. Secondary Outcome: Percentage of Participants With Severity Grade 3 or Above Treatment-Emergent Laboratory Abnormalities
Description: Treatment-emergent laboratory abnormalities were graded using Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 of Adverse Events and Laboratory abnormalities. Laboratory abnormalities were graded as Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe), Grade 4 (Life-threatening), Grade 5 (Death). Percentage of participants with Grade 3 or higher treatment-emergent laboratory abnormalities were reported.
Time Frame: Sequence AB: First dose up to 47 days, Sequence BA: First dose up to 50 days
Population: Participants randomized and received at least 1 dose of that particular study drug with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Atorvastatin | Pravastatin + Rosuvastatin | Filgotinib | Filgotinib + Atorvastatin | Filgotinib + Pravastatin + Rosuvastatin
Number analyzed (Participants) | 26 | 25 | 26 | 24 | 26
percentage of participants | 0 | 0 | 3.8 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events: Sequence AB: First dose up to 47 days, Sequence BA: First dose up to 50 days All Cause-Mortality: Sequence AB: From randomization up to 47 days, Sequence BA: From randomization up to 50 days
Description: Adverse Event: All randomized participants who received at least 1 dose of that particular study drug.
  All Cause-Mortality: All Randomized Analysis Set included all participants randomized into the study after screening.
Arm/Group | Atorvastatin | Pravastatin + Rosuvastatin | Filgotinib | Filgotinib + Atorvastatin | Filgotinib + Pravastatin + Rosuvastatin
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/27 | 0/27 | 0/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/25 | 0/26 | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 2/26 | 4/25 | 13/26 | 2/26 | 0/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Atorvastatin (N=26) | Pravastatin + Rosuvastatin (N=25) | Filgotinib (N=26) | Filgotinib + Atorvastatin (N=26) | Filgotinib + Pravastatin + Rosuvastatin (N=26)
Nausea (Gastrointestinal disorders) | 0 | 1 | 3 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 2 | 8 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2020-09-25): https://cdn.clinicaltrials.gov/large-docs/44/NCT04608344/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-23): https://cdn.clinicaltrials.gov/large-docs/44/NCT04608344/SAP_001.pdf